CLINICAL TRIAL: NCT01367483
Title: An Open-Label, Phase I, Single Dose Study of the Pharmacokinetics, Mass Balance and Disposition of Intravenously Administered 14C-Methylnaltrexone in Normal, Healthy Volunteers
Brief Title: Study of the Pharmacokinetics of Intravenous Administered 14C-MNTX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 102
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1 (Experimental): MNTX active treatment
  Interventions: Drug: IV methylnaltrexone (MNTX)

INTERVENTIONS:
Drug: IV methylnaltrexone (MNTX)

SUMMARY:
This is an open-label, radiotracer study, to be conducted in healthy, normal, male volunteers. It will entail intravenous administration of a single dose of 14C-MNTX, collection of excretions, and periodic drawing of blood samples. Exhaled 14CO2 will also be sampled as a measure of the extent of possible metabolic MNTX demethylation.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 18-45
2. Subject weight between 70 and 90 kg
3. In good physical health, with no evidence at screening of acute or chronic disease likely to affect the investigation

Exclusion Criteria:

1. History or evidence of cardiovascular, gastrointestinal, hepatic, neurological, pulmonary, renal, or other significant chronic condition.
2. Consumption of barbiturates or other inducers or inhibitors of CYP450 isoforms
3. History of or predisposition to erratic or abnormal bowel function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma and Whole Blood Concentration (Cmax) of IV MNTX | 5.5 days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.

SECONDARY OUTCOMES:
Time to Maximum (Tmax) in Plasma and Whole Blood Concentration of IV MNTX | 5.5 Days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.
Clearance of IV MNTX | 5.5 days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.
Half-life of IV MNTX | 5.5 days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.
Volume of Distribution of IV MNTX | 5.5 days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.
Urinary Clearance of IV MNTX | 5.5 days
  To study the pharmacokinetics of MNTX following a single IV dose of 14C-MNTX in normal, healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States